CLINICAL TRIAL: NCT01383460
Title: Randomized Placebo-controlled Trial to Assess the Efficacy of Granulocyte Colony-stimulating Factor (G-CSF) and Erythropoetin (EPO) in the Survival of Patients With Acute-on-chronic Liver Failure (ACLF)
Brief Title: Efficacy of Granulocyte Colony-stimulating Factor and Erythropoetin for Patients With Acute-on-chronic Liver Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS ACLF 01
Record Dates: First submitted 2011-06-26; First posted 2011-06-28 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2012-07

CONDITIONS: Acute on Chronic Hepatic Failure
Keywords: Acute-on-chronic liver failure; ACLF; cirrhosis; acute hepatitis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Fibrosis | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF+EPO (Active Comparator)
  Interventions: Drug: Granulocyte Colony-stimulating Factor (G-CSF) and Erythropoetin (EPO)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Granulocyte Colony-stimulating Factor (G-CSF) and Erythropoetin (EPO) — G-CSF (in prefilled syringe) at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Darbopoetin alpha 100 mcg/ week (in prefilled syringe) for 4 weeks (total 4 doses).
  Arms: G-CSF+EPO
Drug: Placebo — Placebo 1 (in prefilled syringe) s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Placebo 2 every week (in prefilled syringe) for 4 weeks (total 4 doses).
  Arms: Placebo

SUMMARY:
50 patients of Acute-on-chronic liver failure (ACLF) will be enrolled and randomized into G-CSF+EPO or Placebo arms

Treatment protocol To administer G-CSF (in prefilled syringe) at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Darbopoetin alpha 100 mcg/ week (in prefilled syringe) for 4 weeks (total 4 doses).

Standard medical therapy included as per requirement lactulose, bowel wash, albumin, terlipressin, antibiotics (if indicated) will be continued and recorded. Pentoxiphylline in alcoholic hepatitis and Tenofovir in Hep B reactivation Controls: Standard medical therapy will be given along with placebo in similar prefilled syringes.

Follow up Physical examination will be done daily, after 1 week and at 4 weeks, at 2 months, at 3 months and at 6 months CBC on alternate day for 1 week, at end of 1 week and then at end of 4 weeks , at 2 months, at 3 months and at 6 months

KFT on alternate day for 1 week, at end of 1 week and then at end of 4 weeks, at 2 months, at 3 months and at 6 months LFT along with PT/INR on alternate day for 1 week, at end of 1 week and then at end of 4 weeks, at 2 months, at 3 months and at 6 months AFP at baseline, after 4 weeks, at 3 months and at 6 months Liver regenerative potential efficacy testing at baseline and after 4 weeks

DETAILED DESCRIPTION:
50 patients of ACLF will be enrolled and randomized into G-CSF+EPO or Placebo arms

Baseline investigations:

* Hematology

  * CBC, Prothrombin time and INR
  * Peripheral smear, Retics
* Biochemistry

  * Liver function testing, AFP
  * Kidney function test
* Etiology of acute event:

  * Infectious etiology: IgM anti HAV, IgM anti HEV, IgM anti HBc ( If HBsAg +ve), IgM anti HDV ( If HBsAg +ve), HEV RNA
  * Non Infectious etiology: Alcohol binging in last 4 weeks, hepatotoxic drugs, ANA (>1: 80), IgG , surgeries in past 4 weeks, acute variceal bleed within 4 weeks
* Etiology of underlying chronic liver disease :

  * Infectious etiology: total antiHBc, anti HCV, HCV RNA, HBV DNA
  * Non infectious etiology: Autoimmune markers, copper studies, iron studies, HOMA IR, FBS Ascitic fluid analysis ( wherever its possible) UGI endoscopy Imaging USG abdomen with Doppler for spleno-portal axis CECT- Triple phase upper abdomen Liver regenerative potential efficacy testing (wherever it is possible) Histology ( by transjugular liver biopsy) Liver Dendritic cells ( CD11c, CD40, CD 54, CD 123, BDCA 2 staining) by flow cytometry CD 34+ cells and CD 133+ cells measurement in hepatic venous blood, peripheral blood and liver biopsy by flow cytometry Markers of proliferation like ki- 67, proliferating cell nuclear antigen (PCNA) in hepatic venous blood and liver biopsy Markers of angiogenesis like VEGF, v WF in hepatic venous blood Measurement of Hepatic venous pressure gradient ( HVPG)

Treatment protocol To administer G-CSF (in prefilled syringe) at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses), along with Darbopoetin alpha 100 mcg/ week (in prefilled syringe) for 4 weeks (total 4 doses).

Standard medical therapy included as per requirement lactulose, bowel wash, albumin, terlipressin, antibiotics (if indicated) will be continued and recorded. Pentoxiphylline in alcoholic hepatitis and Tenofovir in Hep B reactivation Controls: Standard medical therapy will be given along with placebo in similar prefilled syringes.

Follow up Physical examination will be done daily, after 1 week and at 4 weeks, at 2 months, at 3 months and at 6 months CBC on alternate day for 1 week, at end of 1 week and then at end of 4 weeks , at 2 months, at 3 months and at 6 months

KFT on alternate day for 1 week, at end of 1 week and then at end of 4 weeks, at 2 months, at 3 months and at 6 months LFT along with PT/INR on alternate day for 1 week, at end of 1 week and then at end of 4 weeks, at 2 months, at 3 months and at 6 months AFP at baseline, after 4 weeks, at 3 months and at 6 months Liver regenerative potential efficacy testing at baseline and after 4 weeks

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with acute hepatic insult manifesting as jaundice (Sr. Bil. ≥ 5 mg/dL) and coagulopathy (INR≥1.5), complicated within 4 weeks by ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease

Exclusion Criteria:

* Age <12 or > 75 years
* Autoimmune disorders
* HCC
* Sepsis ( Any culture positive: blood, urine, any other obvious source of infection: UTI, SBP)
* Multi organ failure
* Grade 4 HE
* HIV seropositivity / pregnancy
* Essential Hypertension
* Patients being taken up for transplant
* Refusal to participate in the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Transplant free survival at 3 months. | 3 months

SECONDARY OUTCOMES:
Transplant free survival at 6 months, histo-pathological evidence of hepatic regeneration and mobilization of CD34/stem cells, improvement in severity assessment indices | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, MD, DM, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India